CLINICAL TRIAL: NCT01640054
Title: (OSKIRA-Asia-1X): A Long-term Study to Assess the Safety of Fostamatinib in the Treatment of Rheumatoid Arthritis in Asia
Brief Title: A Long Term Study to Assess the Safety of Fostamatinib in Patients in Asia With Rheumatoid Arthritis
Acronym: OSKIRA-Asia-1X
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AZ decision to discontinue fostamatinib development in RA; rights to fostamatinib returned to Rigel Pharmaceuticals.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4300C00029
Record Dates: First submitted 2012-07-02; First posted 2012-07-13 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dosing regimen (Experimental): Open label Oral treatment 100mg once daily
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib 100mg once daily

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of fostamatinib in patients in Asia with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
(OSKIRA-Asia-1X): A Long-term Study to Assess the Safety of Fostamatinib in the Treatment of Rheumatoid Arthritis in Asia

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures.
* Patients who have successfully completed study D4300C00008 and whose disease is adequately controlled, in the opinion of the Investigator.

Exclusion Criteria:

* Premature withdrawal from study D4300C00008 or in the opinion of the Investigator the patient's disease is not adequately controlled on current treatment.
* Development of any of the withdrawal criteria from study D4300C00008
* Females who are pregnant or breast feeding
* Any other clinically significant disease or disorder, which in the opinion of the Investigator might put the patient at risk due to participation in the study, or may influence the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil - MacKillop, MD, Study Director — AstraZeneca
Locations (26):
- Hong Kong (2):
  - Research Site, Hong Kong, Shatin
  - Research Site, Hong Kong
- Japan (13):
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kato-shi, Hyōgo
  - Research Site, Sendai, Miyagi
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Omura-shi, Nagasaki
  - Research Site, Sasebo-shi, Nagasaki
  - Research Site, Okayama, Okayama-ken
  - Research Site, Tomigusuku-shi, Okinawa
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
- South Korea (4):
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Singapore, Singapore
  - Research Site, Bangkok
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Tanaka Y, Millson D, Iwata S, Nakayamada S. Safety and efficacy of fostamatinib in rheumatoid arthritis patients with an inadequate response to methotrexate in phase II OSKIRA-ASIA-1 and OSKIRA-ASIA-1X study. Rheumatology (Oxford). 2021 Jun 18;60(6):2884-2895. doi: 10.1093/rheumatology/keaa732. PMID 33254235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 115 patients were enrolled; all received at least 1 dose of investigational product. This was an open-label study.
Pre-assignment Details: No patients failed screening.
Groups:
- FOSTA 100 MG QD PO: Fostamatinib 100 mg qd
Period: Overall Study
Arm/Group | FOSTA 100 MG QD PO
Started | 115 (Patients who received treatment)
Did Not Receive Treatment | 0
Completed | 109 (Number of patients on treatment when the study was stopped.)
Not Completed | 6
Not completed — Study-specific disc criteria | 1
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | FOSTA 100 MG QD PO
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 0
  Black or African American | 0
  Asian | 115
  American Indian or Alaska Native | 0
  Indian or Pakistani | 0
  Native Hawaiian or other Pacific Islander | 0

OUTCOME MEASURES:

1. Secondary Outcome: Components of ACR Response Criteria Over Time
Description: ACR = American College of Rheumatology, n/a = not applicable, PO = orally, QD = once daily
Time Frame: Every 12 weeks for one year then every 24 weeks until study end
Population: Insufficient data were available for analysis due to sparse data collection and the early termination of the study.
Arm/Group | FOSTA 100 MG QD PO
Number analyzed (Participants) | 0

2. Secondary Outcome: DAS28-CRP Score Over Time
Description: CRP = C-reactive protein, DAS28 = disease activity score based on a 28 joint count, n/a = not applicable, PO = orally, QD = once daily
Time Frame: Every 12 weeks for one year then every 24 weeks until study end
Population: Insufficient data were available for analysis due to sparse data collection and the early termination of the study.
Arm/Group | FOSTA 100 MG QD PO
Number analyzed (Participants) | 0

3. Secondary Outcome: HAQ-DI Score Over Time
Description: HAQ-DI = health assessment questionnaire - disability index, n/a = not applicable, PO = orally, QD = once daily
Time Frame: Every 12 weeks for one year then every 24 weeks until study end
Population: Insufficient data were available for analysis due to sparse data collection and the early termination of the study.
Arm/Group | FOSTA 100 MG QD PO
Number analyzed (Participants) | 0

4. Secondary Outcome: SF-36 Score Over Time
Description: n/a = not applicable, PO = orally, QD = once daily, SF-36 = 36 item short form health survey
Time Frame: Every 12 weeks for one year then yearly until study end
Population: Insufficient data were available for analysis due to sparse data collection and the early termination of the study.
Arm/Group | FOSTA 100 MG QD PO
Number analyzed (Participants) | 0

5. Primary Outcome: Percentage of Patients Who Had at Least 1 Adverse Event in Any Category
Description: AE = adverse event, IP = investigational product, PO = orally, QD = once daily, SAE = serious adverse event
Time Frame: Entry in extension to study termination (variable duration; maximum 52 weeks)
Population: The full analysis set was the primary population for reporting efficacy and safety data, and comprised all patients who received at least 1 dose of investigational product.
Measure: Number; unit: Percentage of patients
Arm/Group | FOSTA 100 MG QD PO
Number analyzed (Participants) | 115
Percentage of patients
  Any AE | 62.6
  Any AE with outcome of death | 0
  Any SAE (including events with outcome of death) | 3.5
  Any AE leading to discontinuation of IP | 2.6

ADVERSE EVENTS:
Arm/Group | FOSTA 100 MG QD PO
Serious Adverse Events (participants affected / at risk) | 4/115
Other Adverse Events (participants affected / at risk) | 29/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG QD PO (N=115)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG QD PO (N=115)
NEUTROPENIA (Blood and lymphatic system disorders) | 6 (7)
NASOPHARYNGITIS (Infections and infestations) | 14 (18)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (8)
HYPERTENSION (Vascular disorders) | 7 (7)

LIMITATIONS AND CAVEATS:
Insufficient efficacy data was available for analysis due to sparse data collection and the early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days